CLINICAL TRIAL: NCT00386269
Title: Double Blind Randomized Study Into the Efficacy of Codeine Phosphate Analgesia After Cleft Palate Repair in Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Responsible Party: Dr Tracy Assari, Institute of Child Health
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 02AR53
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Cleft Palate Repair
Keywords: codeine phosphate analgesia

INTERVENTIONS:
Drug: Codeine Phosphate Analgesia

SUMMARY:
This study examines the analgesic efficacy of codeine phosphate. It is compared to placebo in infants receiving morphine after surgery. Codeine may be effective enough to make morphine unnecessary.

ELIGIBILITY:
Inclusion Criteria:

* Infants with cleft palate

Ages: 4 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2004-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Dose of morphine used within the first 6h after surgery

SECONDARY OUTCOMES:
Pain scores

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sury, Dr, Principal Investigator — Institute Of Child Health and Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, Anaesthetics, London, United Kingdom